CLINICAL TRIAL: NCT00287716
Title: A Randomized, Double-Blind, Placebo Controlled, Phase 3, Three-Arm Study of the Safety and Efficacy of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Three-Arm Study of the Safety and Efficacy of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIPF-004; Capacity 2
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic; Pulmonary; Fibrosis; Lung; Pirfenidone; InterMune
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2403 mg/day pirfenidone (Active Comparator): Active arm 1, 2403 mg/day pirfenidone dose group.
  Interventions: Drug: Pirfenidone
- 1197 mg/day pirfenidone (Active Comparator): Active arm 2, 1197 mg/day pirfenidone.
  Interventions: Drug: Pirfenidone
- placebo (Placebo Comparator): Placebo equivalent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — 1197 or 2403 mg/day given orally, and administered in divided doses three times daily with food, for the duration of the study.
  Arms: 1197 mg/day pirfenidone; 2403 mg/day pirfenidone
Drug: Placebo — Placebo equivalent, given orally, and administered in divided doses three times daily with food, for the duration of the study.
  Arms: placebo

SUMMARY:
The objectives of this study are to assess the safety and efficacy of treatment with pirfenidone 2403 milligrams per day (mg/d) compared with placebo in patients with idiopathic pulmonary fibrosis (IPF), to assess the safety and efficacy of treatment with pirfenidone 1197 mg/d in patients with idiopathic pulmonary fibrosis and to characterize the pharmacokinetic disposition of pirfenidone in patients with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double blind, placebo-controlled, three-arm, safety and efficacy study of pirfenidone in patients with idiopathic pulmonary fibrosis. Approximately 400 patients at approximately 70 centers will be randomly assigned (2:2:1) to receive either 2403 milligrams (mg) of pirfenidone, placebo equivalent, or 1197 mg of pirfenidone administered in divided doses three times per day (TID) with food. Patients will be randomized by geographic region.

Patients will receive blinded study treatment from the time of randomization until the last patient randomized has been treated for 72 weeks. A Data Monitoring Committee (DMC) will periodically review safety and efficacy data to ensure patient safety.

After week 72, patients who meet the Progression of Disease (POD) definition, which is a ≥ 10% absolute decrease in percent predicted FVC or a ≥ 15% absolute decrease in percent predicted carbon monoxide diffusing capacity (DLco), will be eligible to receive permitted IPF therapies in addition to their blinded study drug. Permitted IPF therapies include corticosteroids, azathioprine, cyclophosphamide and N-acetyl-cysteine (with restrictions).

ELIGIBILITY:
Primary Inclusion criteria:

* diagnosis of idiopathic pulmonary fibrosis
* 40 to 80 years of age
* Forced Vital Capacity greater than or equal to 50% predicted value
* Carbon monoxide diffusing capacity greater than or equal to 35% predicted value
* either Forced Vital Capacity or Carbon monoxide diffusing capacity less than or equal to 90% predicted value
* no improvement in past year
* able to walk 150 meters in 6 minutes and maintain saturation greater than or equal to 83% while on no more than 6 liters per minute (L/min) supplemental oxygen

Primary Exclusion criteria:

* unable to undergo pulmonary function testing
* evidence of significant obstructive lung disease or airway hyper-responsiveness
* in opinion of investigator patient is expected to need and be eligible for a lung transplant within 72 weeks after randomization
* active infection
* liver disease
* cancer or other medical condition likely to result in death within 2 years
* diabetes
* pregnancy or lactation
* substance abuse
* personal or family history of long QT (Q wave,T wave) syndrome
* other IPF treatment
* unable to take study medication
* withdrawal from other IPF trials

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2006-07-14 (Actual); Primary Completion 2008-11-10 (Actual); Study Completion 2008-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- InterMune, Inc., Brisbane, California, United States

REFERENCES:
- [Derived] Behr J, Nathan SD, Costabel U, Albera C, Wuyts WA, Glassberg MK, Haller H Jr, Alvaro G, Gilberg F, Samara K, Lancaster L. Efficacy and Safety of Pirfenidone in Advanced Versus Non-Advanced Idiopathic Pulmonary Fibrosis: Post-Hoc Analysis of Six Clinical Studies. Adv Ther. 2023 Sep;40(9):3937-3955. doi: 10.1007/s12325-023-02565-3. Epub 2023 Jun 30. PMID 37391667
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Kreuter M, Lee JS, Tzouvelekis A, Oldham JM, Molyneaux PL, Weycker D, Atwood M, Kirchgaessler KU, Maher TM. Monocyte Count as a Prognostic Biomarker in Patients with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2021 Jul 1;204(1):74-81. doi: 10.1164/rccm.202003-0669OC. PMID 33434107
- [Derived] Glassberg MK, Nathan SD, Lin CY, Morgenthien EA, Stauffer JL, Chou W, Noble PW. Cardiovascular Risks, Bleeding Risks, and Clinical Events from 3 Phase III Trials of Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis. Adv Ther. 2019 Oct;36(10):2910-2926. doi: 10.1007/s12325-019-01052-y. Epub 2019 Aug 10. PMID 31401786
- [Derived] Nathan SD, Costabel U, Albera C, Behr J, Wuyts WA, Kirchgaessler KU, Stauffer JL, Morgenthien E, Chou W, Limb SL, Noble PW. Pirfenidone in patients with idiopathic pulmonary fibrosis and more advanced lung function impairment. Respir Med. 2019 Jul;153:44-51. doi: 10.1016/j.rmed.2019.04.016. Epub 2019 Apr 24. PMID 31153107
- [Derived] Kreuter M, Lederer DJ, Molina-Molina M, Noth I, Valenzuela C, Frankenstein L, Weycker D, Atwood M, Kirchgaessler KU, Cottin V. Association of Angiotensin Modulators With the Course of Idiopathic Pulmonary Fibrosis. Chest. 2019 Oct;156(4):706-714. doi: 10.1016/j.chest.2019.04.015. Epub 2019 Apr 29. PMID 31047956
- [Derived] Nathan SD, Costabel U, Glaspole I, Glassberg MK, Lancaster LH, Lederer DJ, Pereira CA, Trzaskoma B, Morgenthien EA, Limb SL, Wells AU. Efficacy of Pirfenidone in the Context of Multiple Disease Progression Events in Patients With Idiopathic Pulmonary Fibrosis. Chest. 2019 Apr;155(4):712-719. doi: 10.1016/j.chest.2018.11.008. Epub 2018 Nov 22. PMID 30472023
- [Derived] Nathan SD, Lancaster LH, Albera C, Glassberg MK, Swigris JJ, Gilberg F, Kirchgaessler KU, Limb SL, Petzinger U, Noble PW. Dose modification and dose intensity during treatment with pirfenidone: analysis of pooled data from three multinational phase III trials. BMJ Open Respir Res. 2018 Aug 2;5(1):e000323. doi: 10.1136/bmjresp-2018-000323. eCollection 2018. PMID 30116539
- [Derived] Neighbors M, Cabanski CR, Ramalingam TR, Sheng XR, Tew GW, Gu C, Jia G, Peng K, Ray JM, Ley B, Wolters PJ, Collard HR, Arron JR. Prognostic and predictive biomarkers for patients with idiopathic pulmonary fibrosis treated with pirfenidone: post-hoc assessment of the CAPACITY and ASCEND trials. Lancet Respir Med. 2018 Aug;6(8):615-626. doi: 10.1016/S2213-2600(18)30185-1. Epub 2018 Jun 29. PMID 30072107
- [Derived] Paterniti MO, Bi Y, Rekic D, Wang Y, Karimi-Shah BA, Chowdhury BA. Acute Exacerbation and Decline in Forced Vital Capacity Are Associated with Increased Mortality in Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2017 Sep;14(9):1395-1402. doi: 10.1513/AnnalsATS.201606-458OC. PMID 28388260
- [Derived] Kreuter M, Bonella F, Maher TM, Costabel U, Spagnolo P, Weycker D, Kirchgaessler KU, Kolb M. Effect of statins on disease-related outcomes in patients with idiopathic pulmonary fibrosis. Thorax. 2017 Feb;72(2):148-153. doi: 10.1136/thoraxjnl-2016-208819. Epub 2016 Oct 5. PMID 27708114
- [Derived] Nathan SD, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, Glasscock KF, King TE Jr, Lancaster L, Lederer DJ, Lin Z, Pereira CA, Swigris JJ, Valeyre D, Noble PW, Wells AU. Effect of continued treatment with pirfenidone following clinically meaningful declines in forced vital capacity: analysis of data from three phase 3 trials in patients with idiopathic pulmonary fibrosis. Thorax. 2016 May;71(5):429-35. doi: 10.1136/thoraxjnl-2015-207011. Epub 2016 Mar 11. PMID 26968970
- [Derived] Lancaster L, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, King TE Jr, Lederer DJ, Lin Z, Nathan SD, Pereira CA, Swigris JJ, Valeyre D, Noble PW. Safety of pirfenidone in patients with idiopathic pulmonary fibrosis: integrated analysis of cumulative data from 5 clinical trials. BMJ Open Respir Res. 2016 Jan 12;3(1):e000105. doi: 10.1136/bmjresp-2015-000105. eCollection 2016. PMID 26835133
- [Derived] Noble PW, Albera C, Bradford WZ, Costabel U, Glassberg MK, Kardatzke D, King TE Jr, Lancaster L, Sahn SA, Szwarcberg J, Valeyre D, du Bois RM; CAPACITY Study Group. Pirfenidone in patients with idiopathic pulmonary fibrosis (CAPACITY): two randomised trials. Lancet. 2011 May 21;377(9779):1760-9. doi: 10.1016/S0140-6736(11)60405-4. Epub 2011 May 13. PMID 21571362

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirfenidone 2403 mg/Day: pirfenidone, total daily dose of 2403 mg/day, given as 3 divided doses 3 times/day
- Pirfenidone 1197 mg/Day: pirfenidone, total daily dose of 1197 mg/day, given as 3 divided doses 3 times/day
- Placebo: placebo equivalent, given as 3 divided doses 3 times/day
Period: Overall Study
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Started | 174 | 87 | 174
Completed | 136 | 70 | 143
Not Completed | 38 | 17 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo | Total
Number analyzed (Participants) | 174 | 87 | 174 | 435
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 28 | 73 | 176
  >=65 years | 99 | 59 | 101 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.15) | 68 (7.63) | 66.3 (7.53) | 66.4 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 22 | 46 | 124
  Male | 118 | 65 | 128 | 311
Region of Enrollment [Number; unit: participants]
  United States | 114 | 58 | 114 | 286
  Europe | 34 | 18 | 38 | 90
  Mexico | 2 | 0 | 1 | 3
  Canada | 21 | 8 | 18 | 47
  Australia | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Secondary Outcome: Categorical Assessment of Absolute Change in Percent Predicted Forced Vital Capacity (FVC)
Description: Based on the change in baseline percent predicted FVC at week 72, patients were assigned to 1 of 5 categories: mild decline (<10% but >=0% decline), moderate decline (<20% but >=10% decline), severe decline (>=20% decline), mild improvement (>0% but <10% improvement), or moderate improvement (>=10% improvement). Those who died or had a lung transplant before Week 72 were included in the severe decline category. The results indicate the number of patients who experienced a Categorical Change in Percent Predicted Forced Vital Capacity.
Time Frame: baseline up to 72 weeks
Measure: Number; unit: Patients
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Patients
  Severe decline of >=20%, death, or lung transplant | 14 | 9 | 27
  Moderate decline of <20% but >=10% | 21 | 14 | 33
  Mild decline of <10% but >=0% | 97 | 51 | 90
  Mild improvement of >0% but <10% | 40 | 12 | 24
  Moderate improvement of >=10% | 2 | 1 | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined as the first occurrence of a 10% absolute decline from baseline in percent predicted Forced Vital Capacity, a 15% absolute decline from baseline in percent predicted hemoglobin(Hgb)-corrected carbon monoxide diffusing capacity (DLco), or, death.
Time Frame: Baseline to Week 72
Measure: Number; unit: Number of Patients with Progression
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Number of Patients with Progression
  Death or Disease Progression | 45 | 28 | 62
  Decline in Percent Predicted FVC >=10% | 28 | 16 | 39
  Decline in Percent Predicted DLco >=15% | 9 | 5 | 9
  Death Before Disease Progression | 8 | 7 | 14
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/Day vs Placebo; The null hypothesis is that there is no treatment difference between the pirfenidone 2403 mg/day treatment group and the placebo treatment group; Test type: Superiority or Other; p = 0.023, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.44 to 0.95]

3. Secondary Outcome: Change in Six-Minute Walk Test (6MWT)Distance
Description: The change from Baseline to week 72 in distance walked during the 6-Minute Walk Test as measured in meters (m).
Time Frame: Baseline to Week 72
Measure: Mean (Standard Deviation); unit: Change in Distance Walked in Meters
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Change in Distance Walked in Meters | -60 (121) | -76 (132) | -77 (135)

4. Secondary Outcome: Change in Worst Oxygen Saturation by Pulse Oximetry (SpO2) Measurement Observed During the 6-Minute Walk Test
Description: The change from baseline to week 72 in worst oxygen saturation during the 6-Minute Walk Test as measure by Pulse Oximetry (SpO2) Level is calculated as the simple difference between baseline SpO2 measurements and week 72 SpO2 measurements.
Time Frame: Baseline to Week 72
Measure: Mean (Standard Deviation); unit: Change,Worst Oxygen Saturation (Percent)
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Change,Worst Oxygen Saturation (Percent) | -2 (4) | -1 (5) | -2 (5)

5. Secondary Outcome: Change in Percent Predicted Hemoglobin (Hb)-Corrected Carbon Monoxide Diffusing Capacity (DLco) of the Lungs
Time Frame: Baseline to Week 72
Measure: Mean (Standard Deviation); unit: Change in Percent Predicted DLco
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Change in Percent Predicted DLco | -8 (10) | -9 (11) | -10 (12)

6. Primary Outcome: Absolute Change in Percent Predicted Forced Vital Capacity (FVC)
Description: Mean Change in Percent Predicted Forced Vital Capacity (FVC) as measured from baseline to week 72.
Time Frame: From baseline up to 72 weeks
Measure: Mean (Standard Deviation); unit: Change in Percent Predicted FVC
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Change in Percent Predicted FVC | -8.0 (16.47) | -10.0 (16.68) | -12.4 (18.45)

7. Secondary Outcome: Change in Dyspnea Score
Description: The mean change from baseline to week 72 in Dyspnea score was measured by the University of San Diego Shortness of Breath Questionnaire (UCSD SOBQ). The SOBQ is used to assess shortness of breath with various activities of daily living (for example, brushing ones teeth or mowing the lawn). Patients rated the severity of their shortness of breath experienced on an average day during the past week on a 6 point scale (0 to 5), with 0 = not at all breathless, 4= severely breathless and 5 = Maximally or unable to do because of breathlessness.
Time Frame: Baseline to Week 72
Measure: Mean (Standard Deviation); unit: Change in Dyspnea Score
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Change in Dyspnea Score | 12 (24) | 14 (25) | 15 (26)

8. Secondary Outcome: Worsening of Idiopathic Pulmonary Fibrosis (IPF)
Description: Worsening of IPF was defined by the occurrence of any of the following events:
  Acute IPF exacerbation, IPF-related death, Lung transplantation, or Respiratory hospitalization.
Time Frame: Time to acute IPF exacerbation, IPF-related death, lung transplant or respiratory hospitalization, whichever comes first.
Measure: Number; unit: Number of Patients Who Worsened
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Number analyzed (Participants) | 174 | 87 | 174
Number of Patients Who Worsened | 26 | 10 | 30
Statistical Analysis 1: Comparison: Pirfenidone 2403 mg/Day vs Placebo; The null hypothesis is that there is no treatment difference between the pirfenidone 2403-mg/d treatment group and the placebo treatment group; Test type: Superiority or Other; p = 0.515, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.50 to 1.42]

ADVERSE EVENTS:
Arm/Group | Pirfenidone 2403 mg/Day | Pirfenidone 1197 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 60/174 | 28/87 | 58/174
Other Adverse Events (participants affected / at risk) | 171/174 | 86/87 | 169/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone 2403 mg/Day (N=174) | Pirfenidone 1197 mg/Day (N=87) | Placebo (N=174)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhagic Disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Angina Pectoris (Cardiac disorders) | 2 | 2 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 3 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0
COR Pulmonale Acute (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 3 | 2
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0 | 0
Hypertrophic Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2 | 4
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Right Ventricular Failure (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0
Eye Haemorrhage (Eye disorders) | 0 | 1 | 1
Maculopathy (Eye disorders) | 0 | 1 | 0
Retinal Vein Occulusion (Eye disorders) | 0 | 0 | 1
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colonic Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Erosive Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 0 | 1
Internal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Localised Intraabdominal Fluid Correction (Gastrointestinal disorders) | 0 | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1 | 1
Chest Pain (General disorders) | 5 | 3 | 3
Fatigue (General disorders) | 0 | 0 | 1
Impaired Healing (General disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 2
Oedema Peripheral (General disorders) | 0 | 1 | 0
Vestibulitis (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 2
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal Wall Infection (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Empyema (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0
Lobar Pneumonia (Infections and infestations) | 2 | 2 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1
Perianal Abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 3 | 6
Pneumonia Primary Atypical (Infections and infestations) | 0 | 0 | 1
Post Procedural Infection (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection Fungal (Infections and infestations) | 0 | 1 | 0
Vulval Abscess (Infections and infestations) | 1 | 0 | 0
Burns First Degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns Second Degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post Procedural Myocardial Infarction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood Amylase Increased (Investigations) | 0 | 0 | 1
Gamma-Glutamyltransferase Increasesd (Investigations) | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anoxic Encephalopathy (Nervous system disorders) | 0 | 1 | 0
carotid Artery Stenosis (Nervous system disorders) | 0 | 1 | 1
Cerebral Artery Occlusion (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Migraine with Aura (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 1 | 1
Thrombotic Stroke (Nervous system disorders) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 2 | 0
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urethral Disorder (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 13 | 5 | 14
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Orthostatic Hypertension (Vascular disorders) | 0 | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone 2403 mg/Day (N=174) | Pirfenidone 1197 mg/Day (N=87) | Placebo (N=174)
Abdominal distension (Gastrointestinal disorders) | 15 (16) | 3 (3) | 12 (14)
Abdominal pain (Gastrointestinal disorders) | 16 (18) | 6 (7) | 7 (10)
Anorexia (Metabolism and nutrition disorders) | 19 (20) | 9 (11) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (28) | 9 (10) | 13 (15)
Asthenia (Gastrointestinal disorders) | 15 (18) | 10 (11) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 17 (18) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 33 (42) | 14 (18) | 17 (19)
Dyspepsia (Gastrointestinal disorders) | 30 (34) | 12 (17) | 16 (34)
Hot flush (Vascular disorders) | 11 (11) | 3 (3) | 2 (3)
Insomnia (Psychiatric disorders) | 22 (27) | 13 (14) | 12 (13)
Nausea (Gastrointestinal disorders) | 60 (96) | 22 (27) | 32 (37)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 2 (2) | 5 (9)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 25 (40) | 6 (6) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (15) | 5 (8) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 53 (75) | 15 (27) | 18 (25)
Stomach discomfort (Gastrointestinal disorders) | 14 (16) | 4 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 24 (34) | 11 (14) | 7 (9)
Weight decreased (Investigations) | 15 (15) | 8 (8) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other